CLINICAL TRIAL: NCT06834828
Title: Prevalence of Cusp Asymmetry , Coronary Ostial Eccentricity in Patients Undergoing Trans Catheter Aortic Valve Implantation and Their Impact on Coronary Ostial OverlaP Risk Assessment: an Egyptian CO-OPRA Cohort Study
Brief Title: Prevalence of Cusp Asymmetry, Coronary Ostial Eccentricity in Patients Undergoing Trans Catheter Aortic Valve Implantation and Their Impact on Coronary Ostia Overlap Risk Assessment
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD140/2023
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2023-07

CONDITIONS: Severe Aortic Stenosis; Trans-catheter Aortic Valve Implantation; Coronary Ostial Eccentricity
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe Aortic stenosis patients underwent trans catheter Aortic valve Implantation

SUMMARY:
The goal of this observational study is to measure the prevalence of Cusps asymmetry, coronary Ostial eccentricity in patients with severe aortic stenosis undergoing Trans-catheter Aortic Valve Implantation (TAVI) and measure the degree of coronary ostia overlap with trans-catheter neo-commissure. The main question it aims to answer is:

Do coronary ostial eccentricity or cusp asymmetry have impact on coronary ostia overlap with trans-catheter neo-commissure? Participants already taking TAVI as part of their regular medical care for severe symptomatic aortic stenosis will do post procedural ECG-gated non contrast Multi-detector Computed Tomographic Angiography (MDCTA).

DETAILED DESCRIPTION:
All patients will be subjected to:

Pre-procedural data:

1. Proper history taking including:

   * Age.
   * Sex
   * Body weight, height, and calculated body mass index
   * Previous related medical history (Hypertensive, Diabetic, Rheumatic heart disease, Peripheral vascular disease, Cerebrovascular disease, Chronic kidney disease, Chronic lung disease.)
   * Previous coronary artery disease (completely revascularized or non-revascularized)
   * Previous related surgical history (Surgical valve replacement, Coronary artery bypass graft surgery (CABG) or PCI, Peripheral vascular stenting or bypass graft surgery and carotid stenting or endarterectomy).
2. 12-lead surface electrocardiogram (ECG):

   * Intrinsic rhythm.
   * PR interval duration.
   * QRS duration.
   * Presence or absence of bundle branch block.
   * Baseline ischemic ECG changes (Q waves, ST segment depression or elevation and T wave inverted or flat).
3. Transthoracic echocardiography:

   * Left Ventricular (LV) internal dimensions (end diastolic and end systolic)
   * LV wall thickness and symmetricity (septum and posterior wall)
   * LV ejection fraction by M- mode and 2D eye balling.
   * Resting segmental LV wall motion abnormality.
   * Peak and mean pressure gradient across AV.
   * AV area using continuity.
   * AV leaflets number (tricuspid or bicuspid), thickening and degree of calcification.
   * Presence or absence and degree of Aortic regurgitation (AR).
   * Mitral valve annulus calcification.
   * Presence or absence of Mitral valve regurgitation.
4. Multi-detector Computed Tomographic Angiography (MDCTA) using pre-TAVI protocol:

Pre-procedural contrast enhanced MD cardiac CT imaging will be performed in all patients, Image acquisition will be performed with electrocardiographic gating. All CT data will be reconstructed using images in systolic phase (25-35%) intervals throughout the cardiac cycle with a slice thickness and a slice increment of 0.5 mm and will be analyzed using Osirix viewer software.

All the following parameter and data will be collected pre-procedural:

* Calcium score of aortic annulus and degree of valve calcification and calcium distribution
* LV outflow tract (LVOT) calcification
* Aortic annulus (mean diameters, area derived diameter, perimeter derived diameter)
* Diameter of sinus of Valsalva.
* Height of coronary ostia.
* Assessment of coronary arteries (calcification, degree of plaque causing stenosis, plaque type, presence of previously deployed stents regarding site and their patency if feasible, and the need for pre-TAVI invasive selective coronary angiography with or without PCI).
* Assessment of arterial access (minimal lumen diameter, tortuosity, and calcium distribution).
* Assessment of cusp symmetry:

After identifying the aortic annulus on cardiac CT imaging, a parallel plane few millimeters above the aortic annulus, where all 3 commissures are clearly visible, will be used to evaluate cusp symmetry.

The angle between both commissures of each cusp will be measured and the largest cusp will be identified and classified into 4 categories according to the angle of the largest cusp.

1. Symmetric (120°-125°)
2. Mildly asymmetric (125°-130°)
3. Moderately asymmetric (130°-135°)
4. Severely asymmetric (> 135°). - Assessment of Coronary ostia eccentricity:

Based on the angle deviation between each coronary ostium and the bisector of the corresponding cusp, the eccentricity of coronary ostia will be classified as:

1. Centered (0°-10°).
2. Mildly eccentric (10-20°).
3. Moderately eccentric (20°-30°).
4. Severely eccentric (>30°)

   * Coplanar view by using nadir of each cusp at level of annulus.
   * Cusp Overlap view by overlapping nadirs of right coronary cusp (RCC) and left coronary cusp (LCC)
   * Coronary ostia overlap view using coronary ostium of right coronary artery (RCA) and left coronary artery (LCA) instead of the nadirs of RCC and LCC respectively also at level of annulus, then measuring the difference between two angles in LAO/RAO and Cranial /caudal projection.
   * The angular difference between the right/left cusp and coronary ostia overlap view will be calculated by subtracting the latter fluoroscopic angulation from the prior angulation in both right anterior oblique (RAO)/left anterior oblique (RAO/LAO) and caudal/cranial coordinates. Scatterplots will be composed with RAO/LAO angles at the x-axis and cranial/caudal angles at the y-axis, to show the spatial distribution of both fluoroscopic views and to illustrate the intra-patient fluoroscopic angular difference for every patient.

Post-procedural data:

1. 12-lead surface electrocardiogram (ECG) immediate post procedure and pre discharge:

   * Intrinsic rhythm.
   * PR interval duration.
   * QRS duration.
   * Presence or absence of bundle branch block.
   * Changes indicating ongoing myocardial ischemia (Q waves, ST segment depression or elevation and T wave inverted or flat).
2. Transthoracic echocardiography immediate post procedure and pre-discharge:

   * LV ejection fraction by M- mode and 2D eye balling.
   * Resting segmental LV wall motion abnormality.
   * Peak and mean pressure gradient across implanted AV.
   * Presence of pericardial effusion.
   * Presence of paravalvular leakage (PVL) and PVL degree.
3. ECG gated MDCT post TAVI:

Post-procedural non contrast enhanced MD cardiac CT imaging will be performed in all patients; Image acquisition will be performed with electrocardiographic gating. All CT data will be reconstructed using images in systolic phase (25-35%) intervals throughout the cardiac cycle with a slice thickness and a slice increment of 0.5 mm and will be analyzed using Osirix viewer software.

Based on identification of neo-commissures by commissural markers (CM) (i.e. commissural posts in Acurate neo 2 and C tap in Evolut R /Pro) assessment of coronary overlap (CO) and commissural misalignment (CMA) can be possible as following:

- Coronary overlap (CO): By measuring the angle between each coronary ostium (RCA and LCA) and nearest neo-commissure and categorize CO into 3 groups

1. Severe overlap when < 20°.
2. Moderate overlap when 20-35°.
3. Optimal overlap when > 35°.

ELIGIBILITY:
Inclusion Criteria:

* Severe Aortic stenosis with tri-leaflets aortic valve undergoing Trans catheter Aortic valve Implantation

Exclusion Criteria:

* severe Aortic stenosis with bicuspid leaflets aortic valve
* severe Aortic stenosis undergoing surgical aortic valve replacement

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Severe Aortic stenosis with tri-leaflets aortic valve undergoing Trans catheter Aortic valve Implantation
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Coronary Ostia Overlap with neo-commissures | With in 30 days from indexed procedure
  Measuring angle between trans catheter Aortic valve neo-commissures and coronary Ostia

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University, Abbasia, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
share individual participant data may requires participant approval